CLINICAL TRIAL: NCT05410860
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Etripamil Nasal Spray Self-Administration for the Termination of Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia in Chinese Patients
Brief Title: Efficacy and Safety Study of Etripamil Nasal Spray Self-Administration for the Termination of Spontaneous Episodes of Paroxysmal Supraventricular Tachycardia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Collaborators: Milestone Pharmaceuticals Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JX02002; CTR20221163 (Other: China CDE clinical trial registration)
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-09

CONDITIONS: Tachycardia, Supraventricular; Paroxysmal Supraventricular Tachycardia
Keywords: Etripamil; Paroxysmal supraventricular tachycardia; Cardiac monitoring; Calcium channel blocker; Conversion rate; Chinese patient
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Patients who pass the test dose of the Etripamil NS dosing regimen will be randomized in a 1:1 ratio to Etripamil NS 70mg or placebo using an Interactive Response Technology (IRT) system.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Etripamil NS 70 mg with Optional Second Dose (Experimental): Dosing regimen that permits a second dose of Etripamil NS 70 mg
  Interventions: Drug: Etripamil NS 70 mg
- Placebo with Optional Second Dose (Experimental): Dosing regimen that permits a second dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etripamil NS 70 mg — Etripamil NS 70 mg will be administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Arms: Etripamil NS 70 mg with Optional Second Dose
Drug: Placebo — Placebo will be administered via the Aptar Pharma Nasal Spray Bidose System, supplied as prefilled devices packaged into child-resistant boxes with instructions for use provided in the study drug box.
  Arms: Placebo with Optional Second Dose

SUMMARY:
To determine whether etripamil nasal spray (NS) self-administered by Chinese patients is superior to placebo at terminating episodes of PSVT in an at-home setting； To evaluate the efficacy of etripamil NS self-administered by Chinese patients compared with placebo on a range of clinical markers.

To evaluate the safety of etripamil NS self-administered by Chinese patients compared with placebo

DETAILED DESCRIPTION:
The study is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of etripamil NS self-administered by patients who experience an episode of PSVT in an at-home setting.

This is an event-driven study. Enrollment into the study will continue until the adjudication of the 180th positively adjudicated PSVT episode in patients treated with double-blind study drug during the Randomized Treatment Period required for the study's pivotal analysis. After the date of the adjudication of the 180th positively adjudicated PSVT episode, all randomized patients will be unblinded at this timepoint and enter into an approximately 6 months open-label period of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Male or female patients at least 18 years of age;
2. Electrographically documented history of PSVT (e.g., diagnosis based on ECG , Holter monitoring, etc.). If patient had a prior ablation for PSVT, patient must have documented ECG evidence of PSVT post-ablation;
3. History of sustained episodes of PSVT (i.e., typically lasting 20 minutes or longer);
4. Females of childbearing potential who are sexually active with a male partner who is not surgically sterile (i.e., vasectomy) must agree to use an approved highly effective form of contraception from the time of signed informed consent until 30 days after the last administration of study drug.;

   The following categories define females who are NOT considered to be of childbearing potential:
   * Premenopausal females with 1 of the following:

     1. Documented hysterectomy;
     2. Documented bilateral salpingectomy or tubal ligation; or
     3. Documented bilateral oophorectomy; or
   * Postmenopausal females, defined as having amenorrhea for at least 12 months without an alternative medical cause; and
5. Signed written informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Systolic blood pressure (SBP) <90 mmHg after a 5-minute rest in sitting position at the Screening Visit or before the test dose. In patients treated with a chronic prophylactic drug for PSVT (e.g., beta blockers, verapamil, and diltiazem), the drug may be stopped for at least the equivalent of 5 half-lives, patients may be rescreened once, and chronic use of the drug cannot be restarted after randomization;
2. History of severe symptoms of hypotension, especially syncope, during episodes of PSVT;
3. History of atrial arrhythmia that does not involve the atrioventricular (AV) node as part of the tachycardia circuit (e.g., atrial fibrillation, atrial flutter, intra-atrial tachycardia);
4. History of allergic reaction to verapamil;
5. Current therapy with digoxin or any Class I or III antiarrhythmic drug, except if these drugs are stopped at least the equivalent of 5 half-lives before the Test Dose Randomization Visit;
6. Current chronic therapy with oral amiodarone, or have taken oral amiodarone within 30 days prior to the Test Dose Randomization Visit;
7. Evidence of ventricular pre-excitation (e.g., delta waves, short PR interval <100 msec, Wolff Parkinson White syndrome) on the ECG performed at the Screening Visit or before the test dose administration;
8. Evidence of a second- or third-degree AV block on the ECG performed at the Screening Visit or before the test dose administration;
9. History or evidence of severe ventricular arrhythmia (e.g., torsades de pointes, ventricular fibrillation, or ventricular tachycardia);
10. Current congestive heart failure defined by the New York Heart Association Class II to IV;
11. History of Acute Coronary Syndrome or stroke within 6 months of screening;
12. Evidence of hepatic dysfunction ;
13. Evidence of End-Stage Renal Disease;
14. Females who are pregnant or lactating;
15. Evidence or history of any significant physical or psychiatric condition including drug abuse, which, in the opinion of the Investigator, could jeopardize the safety of patients or affect their participation in the study. Additionally, the Investigator has the ability to exclude a patient if for any reason the Investigator judges the patient is not a good candidate for the study (e.g., illiteracy or poor understanding) or will not be able to follow study procedures;
16. Participation in any investigational drug or device study or the use of any investigational drug or device within 30 days or five terminal phase half-lives of the drug whichever is longer, prior to the Screening Visit; or
17. Previously enrolled in a clinical trial for Etripamil and received study drug during a perceived episode of PSVT;
18. An immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Before randomization in this study, all patients will receive a test dose of an etripamil NS dosing regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Time to an adjudicated termination of a positively adjudicated episode of PSVT and conversion to sinus rhythm (SR) for at least 30 seconds within 30 minutes of start of study drug dosing | Within 30 minutes of start of study drug dosing.
  The primary efficacy endpoint is defined as an adjudicated termination of a positively adjudicated episode of PSVT (AV nodal reentrant tachycardia or AV reentrant tachycardia determination if possible) and conversion to sinus rhythm (SR) for at least 30 seconds within 30 minutes of start of study drug dosing.

SECONDARY OUTCOMES:
Time to conversion at time points of 5, 10, 15, 45, and 60 minutes | 1 hour after administration of study drug
Time to conversion in patients with the option of repeat administration | 1 hour after administration of study drug
The percentage of patients requiring additional medical intervention in emergency department to terminate an episode of PSVT | Up to 2 years
Number of participants with relief of specific symptoms (i.e., heart palpitations, rapid pulse feeling, chest pain, anxiety, shortness of breath, dizziness, and fainting) | 1 hour after administration of study drug
Rating of Treatment Satisfaction Questionnaire for Medication (TSQM). | 1 hour after administration of study drug
  Treatment satisfaction will be analyzed by comparing the Treatment Satisfaction Questionnaire for Medication 9(TSQM-9) score for satisfaction in the 2 treatment groups. The TSQM-9 is composed of 9 questions with responses on a scale of 1 (extremely dissatisfied) to 7 (extremely satisfied). A higher score indicated greater satisfaction with medication.
The percentage of adverse event | Up to 2 years
Number of participants with arrhythmias and conduction disorders detected on surface electrocardiogram（ECG） or cardiac monitoring system (CMS) recordings. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Chen, Study Director — Corxel Pharmaceuticals; Changsheng Ma, Principal Investigator — Beijing Anzhen Hospital
Locations (53):
- China (53):
  - Baotou Central Hospital, Baotou
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Beijing Anzhen Hospital; Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Chui Yang Liu Hospital Affiliated to Tsinghua University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Central Hospital of China Aerospace Corporation, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The Third Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - Changzhou No.2 People's Hospital, Changzhou
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu
  - The First Hospital of Jilin University, Ch’ang-ch’un
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - People's Hospital of Deyang City, Deyang
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First People's Hospital of Hangzhou Linping District, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Huai'an First People's Hospital, Huai'an
  - Huainan First People's Hospital, Huainan
  - Huizhou Municipal Central Hospital, Huizhou
  - Jinan Central Hospital, Jinan
  - Shandong Province Qianfoshan Hospital, Jinan
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Lishui Municipal Central Hospital, Lishui
  - The First Affiliated Hospital of Henan Science and Technology University, Luoyang
  - Mianyang Central Hospital, Mianyang
  - The Nanchang Third Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning
  - The second affiliated Hospital of Guangxi Medical University, Nanning
  - Nanyang Second General Hospital, Nanyang
  - Ningbo First Hospital, Ningbo
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Pudong New Area People's Hospital, Shanghai
  - Shanghai Tongren Hospital, Shanghai
  - Shangrao People's Hospital, Shangrao
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Jiangsu Taizhou People's Hospital, Taizhou
  - Binhai Hospital (Tianjin Fifth Central Hospital), Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - CR and WISCO General Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Xingtai Third Hospital, Xingtai
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu
  - ZiBo Central Hospital, Zibo